CLINICAL TRIAL: NCT01974726
Title: Gas Supply, Demand and Middle Ear Gas Balance -- Project 1, Specific Aim 4, Protocol 3
Brief Title: Gas Supply, Demand and Middle Ear Gas Balance -- Diagnosis of Eustachian Tube Dysfunction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of funding
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Cuneyt M. Alper, Professor of Otolaryngology, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO13040671-3; 2P50DC007667 (NIH)
Record Dates: First submitted 2013-10-22; First posted 2013-11-01 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Eustachian Tube Dysfunction
Keywords: ear; middle ear; Eustachian tube; Eustachian tube dysfunction; Eustachian tube function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- affected, intact tympanic membranes (Other): History of middle-ear disease, ears with no holes/perforations/patent tympanostomy tubes in eardrum
  Interventions: Other: ET Stress test; Other: Sonotubometry; Other: Maneuver Sequence; Other: 9-Step Test; Other: Tubomanometry; Other: Videoendoscopic assessment of ETF
- affected, non-intact tympanic membranes (Other): History of middle-ear disease, ears with hole/perforation/patent tympanostomy tube in eardrum
  Interventions: Other: ET Stress test; Other: Sonotubometry; Other: Forced Response Test (FRT); Other: Inflation Deflation Test (IDT); Other: Maneuver Sequence; Other: Tubomanometry; Other: Videoendoscopic assessment of ETF
- controls, intact tympanic membranes (Other): No history of middle-ear disease, ears with no hole/perforation/patent tympanostomy tube in eardrum
  Interventions: Other: Sonotubometry; Other: Maneuver Sequence; Other: 9-Step Test; Other: Tubomanometry; Other: Videoendoscopic assessment of ETF; Other: Pressure chamber ET test
- controls, non-intact tympanic membranes (Other): No history of middle-ear disease, ears with hole/perforation/patent tympanostomy tube in eardrum
  Interventions: Other: Sonotubometry; Other: Forced Response Test (FRT); Other: Inflation Deflation Test (IDT); Other: Maneuver Sequence; Other: Tubomanometry; Other: Videoendoscopic assessment of ETF

INTERVENTIONS:
Other: ET Stress test — Performed in pressure chamber. For subjects with intact tympanic membranes, chamber pressure increased from ambient to +2500 daPa (+2000 daPa for children). At that pressure and then at down-stepped pressures of 250 daPa/steps to a chamber pressure of -1500 daPa (or a passive ET opening), the subject will swallow to attempt to open the ET as detected by sonotubometry and/or a change in ear canal pressure. ET passive opening and closing pressures will then be determined. In ears with a non-intact tympanic membrane, a small volume probe connected to a pressure transducer will be placed in the ear canals and the procedure repeated with continuous recording of ME pressure. ET opening is recorded as a change in ME pressure toward local ambient.
  Arms: affected, intact tympanic membranes; affected, non-intact tympanic membranes
Other: Sonotubometry — Microphones are placed in the ear canals and covered with ear protectors. A nasal probe placed in one nostril introduces a white noise to the nasopharynx and the subject is asked to swallow. The test system identifies the sound frequency best transmitted through an open ET (if the test is positive, i.e. ET opens) and the procedure is repeated with the nasal sound pressure delivered at that frequency. The probe is then placed in the contralateral nostril and the procedure repeated. The microphone signals from both ear canals are continuously outputted and recorded. A positive ET opening is defined as a 5 dB increase above baseline during any of the 4 swallows and can be semi-quantified as the area under the baseline-adjusted ear canal sound pressure-time curve. The test is designed to measure the presence or absence of muscle-assisted ET openings during swallowing at local ambient pressure.
Other: Forced Response Test (FRT) — The FRT requires a non-intact tympanic membrane and uses an instrument consisting of an ear canal probe coupled serially to a differential pressure transducer, via a valve to a flow sensor and via a second valve to a variable-speed constant-flow pump. The probe is sealed in the ear canal and both valves are opened. The pump is set to deliver a constant flow of 11 ml/min which increases ME pressure to passively open the ET. This is followed by a decrease in ME pressure to steady state pressure and flow conditions. The subject is asked to swallow which either transiently increases (further ET dilation) or decreases (ET constriction) the transET flow. The pump is turned off causing the ET to close at a residual ME pressure. This procedure is repeated at flow rates of 23 and then 46 ml/min.
  Arms: affected, non-intact tympanic membranes; controls, non-intact tympanic membranes
Other: Inflation Deflation Test (IDT) — The IDT requires a non-intact tympanic membrane and uses the FRT instrument. ME pressure is increased to 250 daPa (ref ambient), the valves to the flow sensor and pump closed and the subject is asked to swallow repeatedly at a natural interval while monitoring ME pressure until further swallowing fails to change ME pressure. The procedure is repeated with an applied under-pressure of -250 daPa. The outcome variable is the percent pressure change (%reduction) at test end. The test measures the muscle-assisted tubal openings under minor stress (ME under-pressure) and facilitative (ME over-pressure) conditions, and can detect a patulous/semi-patulous ET by an inability to maintain applied ME over and/or under-pressures between swallows.
  Arms: affected, non-intact tympanic membranes; controls, non-intact tympanic membranes
Other: Maneuver Sequence — The sequence consists of the Toynbee, Valsalva, Sniffing and Continuous Pressure Test (CPT). The test system consists of ear canal and nasal pressure probes. For the Toynbee test the subject pinches both nostrils (without constricting the nasal probe) and swallows; for the Sniffing test, the subject performs a series of forcible sniffs that must achieve a nasopharyngeal pressure of at least -400 daPa; for the Valsalva test the subject pinches both nostrils and forcibly blows against the closed nose to achieve a nasopharyngeal pressure of at least 400 daPa, and for the CPT the subject breathes through his/her mouth in a relaxed manner for 2 minutes.
Other: 9-Step Test — This test requires an intact tympanic membrane. Middle ear (ME) pressure is recorded by tympanometry before and after application of a 300 daPa over-pressure to the ear canal and then before and after application of a 300 daPa under-pressure to the ear canal. Between steps, the subject is asked to swallow in an attempt to open the ET and change ME pressure. A positive test is indicated by a minimum 10 daPa change in ME pressure after a given swallow and excellent muscle-assisted ET opening is indicated by an initial change to a more negative ME pressure after a swallow, followed by a return to 0 daPa, a positive ME pressure and a return to 0 daPa for sequential swallows. The test is designed to measure the presence/absence of active ET openings during swallowing at ambient pressures.
  Arms: affected, intact tympanic membranes; controls, intact tympanic membranes
Other: Tubomanometry — The test system is commercially available and can test ears with and without an intact tympanic membrane. Pressure sensors are inserted bilaterally into the ear canals and sealed. A controlled air-flow is introduced into the nose and nasopharynx and the subject swallows. ET openings are detected as a change in ME pressure measured directly as a pressure pulse in the ear canal for ears with a non-intact tympanic membrane or indirectly as a change in ear canal pressure caused by tympanic membrane displacement in ears with intact tympanic membranes. The outcome is the detection of a pressure change in the ear canal during swallowing which is indicative of a muscle-assisted tubal opening.
Other: Videoendoscopic assessment of ETF — The subject's nose is topically anesthetized and decongested with 4% lidocaine and 0.05% oxymetazoline. If ventilation tubes are present, probes are sealed in the ear canal(s)and a pressure of 200 daPa is applied to the ME(s) to assess ET opening. If tympanic membranes are intact, microphones for sonotubometry are placed in the ear canals. Then, an endoscope attached to a video camera is introduced into the ipsilateral nasal cavity and focused on the ET orifice. For sonotubometry, the sound source probe is placed in the contralateral nostril. The subject is asked to swallow, vocalize and perform a series of mandibular movements. Signals from the video camera and pressure transducer or sonotubometry microphones are continuously recorded. The data are studied to document dilation of the nasopharyngeal ET orifice during swallowing and to rule in or out an anatomical or functional nasopharyngeal abnormality as the cause of a diagnosed ET dysfunction.
Other: Pressure chamber ET test — Performed in pressure chamber. Pressure increased to create middle-ear underpressure, then subject is asked to swallow several times. Middle-ear pressures are then measured by tympanometry. This is repeated with decreased chamber pressure, creating a middle-ear overpressure.
  Arms: controls, intact tympanic membranes

SUMMARY:
The aim of this study is to determine which of the many Eustachian tube function tests (or combination of tests) is most helpful in finding out what is causing ear problems in children and adult patients with middle-ear diseases thought to be due to poor Eustachian tube function. The Eustachian tube is a biological tube that connects the middle ear to the back of the nose and throat. When the Eustachian tube works normally, it opens and closes to help keep the pressure in the middle ear the same as room air-pressure (atmospheric pressure). When the Eustachian tube does not work well, the pressure in the middle ear can increase or decrease and feel like a blocked ear or cause ear pain. Poor Eustachian tube function can be associated with distressing middle-ear symptoms, predispose to middle-ear problems under conditions of rapidly changing air pressures such as occur during airflight and diving, and cause certain middle-ear diseases such as otitis media with effusion. It is also known that the results for the most commonly used Eustachian tube function tests in adults and children with various middle-ear diseases are poorer when compared to children and adults without middle-ear diseases. However, knowing that there is a difference in test results between groups with and without disease does not mean that any of those tests provide information useful in the management of individual patients with diseases due to Eustachian tube function. To be useful clinically, a test(s) that can accurately identify patients with a level of poor Eustachian tube function sufficient to cause middle-ear symptoms and signs and/or cause middle-ear disease is needed. To be very useful, tests should be able to diagnose the cause of any observed Eustachian tube problem so that treatment for that problem could be begun. The investigators would also want tests that could predict whether or not the ear disease will resolve with (or without) treatment and whether or not certain surgical procedures for middle-ear problems will be successful. Here, a number of Eustachian tube function tests are being used to diagnose and characterize the cause of Eustachian tube dysfunction in children and adults presenting to the research clinic with suspected poor Eustachian tube function and/or a recent history of middle-ear disease that can be caused by poor Eustachian tube function. After the testing, medical records will be periodically reviewed for 2 years and study participants will be contacted by phone to obtain information on their middle-ear disease, the response of the disease to any treatments and the success/failure of any surgical procedures used to fix middle-ear problems.

Because this study focuses on evaluating the potential usefulness of Eustachian tube function testing for the diagnosis of Eustachian tube dysfunction and, if present, its cause, no specific treatments or surgical interventions are included in this study or recommended by the investigators. These decisions are left to the subject-patient in consultation with their doctor.

To further evaluate the Eustachian function tests, a control group of healthy adults without a history of middle-ear problems will undergo testing at two separate sessions; these subjects will have no further follow-up.

DETAILED DESCRIPTION:
The overall objective is to develop the clinical utility of a panel of new and existing Eustachian Tube Function (ETF) tests with respect to diagnosing ET dysfunction and its cause, recommending specific targeted interventions to re-establish normal function and predicting the future course of diseases attributable to that dysfunction.

In this Protocol, the investigators open their research center to the clinical evaluation of all physician or self-referred children and adults with suspected ET dysfunction (ETD)and/or diseases attributable to that dysfunction, perform a broad panel of ETF tests to diagnose the presence/absence and cause of the dysfunction and then collect from patient records information on the future disease course in those subjects to begin developing a comprehensive database relevant to clinical utility of the various tests. An adult control group consisting of healthy volunteers without a history of significant middle-ear disease will also be entered.

ETF will be evaluated in this highly heterogeneous population using a pressure-chamber protocol (ET stress test), a panel of other tests as is relevant to the status of the tympanic membrane and, in older subjects (10 years and older, or younger if tolerated), endoscopic assessments of nasopharyngeal pathologies. The goal of this study is to define the least costly panel of test procedures that is sensitive, specific and accurate for the diagnosis of ETD, identification of the cause of the dysfunction if observed, prediction of the success rates for medical or surgical interventions (e.g. the newer ET surgical procedures, adenoidectomy, myringoplasty) and prediction of future disease course (probability of spontaneous resolution). These results will be interpreted in terms of whether or not ETF testing is of practical value to clinicians in their decision-making related to ETD, otitis media with effusion (OME) and chronic OME (COME) and if relatively portable, inexpensive test systems with the listed properties can be introduced into a typical physician's practice.

All entered patients/subjects with a history of middle-ear disease will have an initial history taken with a focus on predisposing factors for ETD and OME (e.g. atopy, recent or frequent colds, gastroesophageal reflux disease, etc.) and on the symptoms and signs associated with the initial presentation of the condition. A standard clinical ear, nose and throat (ENT) examination with pneumatic otoscopy and tympanometry (if possible) will be done. Subjects with extant middle-ear (ME) effusion or otorrhea through a tube or with signs or symptoms of a cold or allergic rhinitis will not be tested, but may be studied at a later time upon resolution of the condition. Patients with no contraindications to the planned test panel will be triaged to one of the two standard ETF test panels used in our laboratory, 1) the Maneuver Sequence, sonotubometry, tubomanometry, the Forced-Response test, the Inflation-Deflation test and the ET stress test if presenting with a tympanic membrane perforation/ventilation tube, or 2) the Maneuver Sequence, sonotubometry, tubomanometry, 9-step test and the the ET stress test if presenting with an intact tympanic membrane. The investigators begin with these tests because they capture a global assessment of ETF with respect to: the muscle-assisted ET opening efficiency which is a measure of ME pressure-regulation and the patency of the ET which is a measure of the protective function of the ET (patulous, semi-patulous, obstructed). For all subjects aged 10 years and older and any younger subject who is sufficiently cooperative, the investigators will perform nasoendoscopic evaluations of the nasopharynx and ET orifice at rest and during swallowing, speech and other maneuvers to determine if there is a detectable extrinsic cause of the ETD. A summary diagnosis of the presence/absence and the type and cause of the ETD (if any) will be prepared by the study physician, and, if a referred patient, submitted to the referring physician or, if self-presenting, to the subject's Primary Care Physician (PCP). Every 6 months for 2 years, the subjects or their parents (if minors) will be contacted to update their medical history, and the subject's medical charts will be requested and reviewed once a year for 2 years to update the Center's database with respect to the subject's disease course and the outcome of any surgeries or treatments.

The adult control subjects will undergo similar ET function testing as the affected group and nasoendoscopic evaluation. These will be repeated at one other test session at least 1 week after the first testing and there will be no further follow-up of these subjects.

Using the control data from parallel studies, the control subjects in this protocol and the subjects' history with respect to ME complaints, the evaluations of ETF, the feedback from subjects and the review of medical records, the investigators expect to develop an algorithm that prescribes the specific test sequences that optimize the diagnosis of the type and cause of ETD and the treatment recommendations for a given patient presenting with a specific history and set of ETD signs and/or symptoms. The investigators also expect to establish, with reasonable certainty, whether or not the results of these tests are clinically useful to otolaryngologists and general practitioners in their decision-making with respect to prescribed treatments and/or surgical interventions for affected patients. For each test or panel of tests, the investigators will define their sensitivity, specificity and accuracy with respect to the various outcomes.

ELIGIBILITY:
AFFECTED SUBJECTS:

Inclusion Criteria:

* 3-70 years of age
* Diagnosed or suspected Eustachian tube dysfunction or middle-ear disease
* Able to read and comprehend English

Exclusion Criteria:

* Extant middle-ear effusion, allergic rhinitis or "cold" (may enter when resolved)
* History of ossicular reconstruction
* Blood pressure greater than or equal to 140/90 (adults)
* Recent angina; history of heart attack, stroke, cardiac surgery or any other medical condition that the study physician deems entry not in the subject's best interest.

CONTROL SUBJECTS

Inclusion Criteria:

* 18 -60 years of age
* Generally healthy
* No history of middle-ear disease
* Intact or non-intact tympanic membrane -- perforation or tube for reasons other than middle-ear disease.

Exclusion Criteria:

* Extant middle-ear effusion, allergic rhinitis or "cold" (may enter when resolved)
* History of ossicular reconstruction
* Blood pressure greater than or equal to 140/90
* Sensitivity to drugs used for endoscopy (lidocaine, oxymetazoline)

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-10; Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
ETF tests | 2 years (affecteds), 1 week (controls)
  sensitivity/specificity of various ETF tests and combinations of tests

CONTACTS AND LOCATIONS:
Overall Officials: Cuneyt M Alper, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Middle Ear Physiology Laboratory, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No